CLINICAL TRIAL: NCT06282146
Title: Testing a Transdiagnostic TMS Treatment Target
Acronym: T5
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joseph J. Taylor, MD, PhD, Instructor in Psychiatry, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024P000252
Record Dates: First submitted 2024-02-06; First posted 2024-02-28 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder; Depression; Psychiatric Disorder; Mood Disorders; Mental Disorder; Anxiety Disorders; OCD; PTSD
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Mental Disorders; Mood Disorders; Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Open-label aiTBS to posterior parietal cortex (Experimental): 10 iTBS treatment sessions per day (18,000 pulses/day) for 5 consecutive days (90,000 pulses total). In the unlikely event that a participant is late for an hourly treatment, then the treatment will be delayed accordingly. The minimum gap between treatments will be 25 minutes. Each iTBS treatment will consist of 60 cycles of 10 bursts of three pulses at 50 Hz delivered in 2-second trains (5 Hz) with an 8-second intertrain interval. Stimulation will be delivered at 90% resting motor threshold (rMT), adjusted for depth of the identified functional connectivity target.
  Interventions: Procedure: transcranial magnetic stimulation

INTERVENTIONS:
Procedure: transcranial magnetic stimulation — non-invasive form of brain stimulation
  Other Names: TMS; accelerated intermittent theta burst stimulation; aiTBS

SUMMARY:
The goal of this clinical trial is to test a new brain stimulation treatment target for individuals with depression plus at least one additional psychiatric disorder. The main question is to understand the safety profile of a non-invasive form of brain stimulation called accelerated intermittent theta burst stimulation when it is targeting the posterior parietal cortex. Additional questions focus on whether this stimulation improves symptoms of depression and other psychiatric disorders as well as whether this stimulation changes brain function.

DETAILED DESCRIPTION:
Psychiatric disorders are often studied individually. However, up to half of individuals who meet criteria for one psychiatric disorder also meet criteria for another. These individuals are difficult to diagnose and treat. Relative to those with one disorder, individuals with two or more have worse treatment outcomes, more functional impairment, and a greater risk of premature death.

Neuromodulation treatments like transcranial magnetic stimulation (TMS) work when routine psychotherapy and medications have not worked, but they typically target one disorder at a time. In fact, the TMS field is largely focused on strategies to make TMS more precise by targeting individual symptoms within a diagnosis. This strategy is important, but it may be difficult to scale and optimize in the setting of real-world psychiatric comorbidity. For example, there are 227 possible ways to meet criteria for major depressive disorder, complicating precision TMS strategies for individuals with or without comorbid disorders.

In this study, the investigators are moving in a different direction by targeting the brain network shared across psychiatric disorders in treatment-seeking individuals with more than one psychiatric disorder. This approach is based upon prior work. In a 2023 Nature Human Behavior study, the investigators analyzed four independent datasets with coordinate and lesion network mapping to test for a brain network shared across psychiatric disorders. They found that atrophy coordinates across six psychiatric disorders (193 studies) mapped to a common brain network defined by positive connectivity to the anterior cingulate and insula, and by negative connectivity to posterior parietal and lateral occipital cortices. The investigators verified that this transdiagnostic network was robust to leave-one-diagnosis-out cross validation and specific to atrophy coordinates from psychiatric versus neurodegenerative disorders (72 studies). Lesion-induced damage to this network correlated with the number of post-lesion psychiatric diagnoses in an independent dataset (194 patients). The transdiagnostic network also aligned with neurosurgical ablation targets for psychiatric disorders (4 targets), suggesting possible therapeutic relevance and generating testable hypotheses for neuromodulation. Importantly, the candidate TMS target that emerges from this transdiagnostic network is also a critical node of the convergent depression network that was derived across 14 independent datasets. This target has not been robustly tested for major depressive disorder (MDD) or transdiagnostic symptoms.

In this open-label pilot trial, the investigators will test the hypothesis that modulating the transdiagnostic network with transcranial magnetic stimulation (TMS) will be safe and tolerable. Secondary outcomes will assess changes in the cumulative burden of psychopathology in individuals with MDD plus at least one additional psychiatric disorder. This approach is novel in three important ways: 1) This study will enroll, not exclude, individuals with multiple psychiatric illnesses. Most clinical trials selectively enroll individuals with a single diagnosis, a strategy that does not generalize to real-world settings where psychiatric comorbidity is common and difficult to treat. 2) The transdiagnostic target was validated with causal sources of information (i.e., brain lesions, neurosurgical ablation). In other words, this study will optimize the "where to stimulate" factor. TMS targets are usually derived from functional neuroimaging studies that identify correlates of illness. These correlates could cause, compensate for, or be epiphenomena of treatment or other variables, an interpretation that matters for TMS. 3) The investigators will use the most rapid-acting and robust TMS protocol. In other words, they will optimize the "how to stimulate" factor. Conventional TMS protocols require scalp-targeted treatments delivered weekdays for 6-8 weeks. By contrast, the accelerated intermittent theta burst (iTBS) protocol in this study is adapted from Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT), which consists of MRI-guided treatment delivered 10 times a day for 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* English proficiency sufficient for informed consent, questionnaires/tasks, and treatment
* Diagnosis of MDD per DSM-5 criteria (Quick Structured Clinical Interview for DSM-5 Disorders) and currently experiencing a moderate to severe episode:
* >20 on Beck Depression Inventory (BDI)
* >20 on the Montgomery-Åsberg Depression Rating Scale (MADRS) 14, 15
* Moderate to severe level of treatment resistance (Maudsley Staging Method)16, 17
* Diagnosis of at least one or more of the following psychiatric conditions per DSM-5 criteria (Quick Structured Clinical Interview for DSM-5 Disorders):
* Generalized anxiety disorder (GAD), panic disorder (PD), or social anxiety disorder (SAD)
* Obsessive compulsive disorder (OCD)
* Post-traumatic stress disorder (PTSD)
* Physician referral for individuals with either schizophrenia or schizoaffective disorder
* Stable psychiatric medication regimen, or remain medication free, for 4 weeks prior to treatment and to remain on this regimen throughout the study until the two-week post-treatment visit
* Primary clinician (e.g. psychiatrist, therapist, psychologist, APRN, PA, etc.) responsible for psychiatric care before, during, and after the trial
* Agreement to lifestyle considerations
* Abstain from becoming pregnant from time of screening to two weeks after treatment (post-treatment MRI visit)
* Continue usual intake patterns of caffeine- or xanthine-containing products (e.g. coffee, tea, soft drinks, chocolate) throughout treatment
* Abstain from alcohol, tobacco, and recreational drugs for at least 24 hours before the start of each MRI and each TMS session

Exclusion Criteria:

* Active pregnancy as determined by a urine pregnancy test
* Positive urine drug screen for illicit substances (not including THC)
* Depressive symptoms refractory to 8 sessions of electroconvulsive therapy (ECT)
* Recent (within 4 weeks) or concurrent use of rapid acting antidepressant agent (ketamine/esketamine/ECT)
* Receiving or planning to receive other TMS treatments during course of participation
* History of
* Autism spectrum disorder
* Neurosurgical intervention for depression
* Intellectual disability
* Severe cognitive impairment
* Significant neurological illness (e.g., dementia, Parkinson's, Huntington's, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis, brain lesion)
* Untreated or insufficiently treated endocrine disorder
* Treatment with investigational drug or intervention during the study period
* Depth-adjusted TMS treatment dose > 65% maximum stimulator output
* Existing tinnitus (ringing in the ears)
* Current evidence of:
* Mania or hypomania
* Active suicidal ideation or a suicide attempt (defined by C-SSRS) within the past year
* Neurological lesion
* Contraindications to either TMS or MRI (e.g., metallic implants, severe insomnia > 4 hours per night with hypnotic, etc.).
* Moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal (not including cannabis or nicotine use disorders)
* Bipolar I disorder
* For participants with schizophrenia or schizoaffective disorder referred by a physician:
* Total PANSS score >90
* Score >4 (moderate-severe) on any positive PANSS item
* Active substance use disorder (other than nicotine)
* Hospitalization for psychosis in the past 6 months
* Severe borderline personality disorder
* Any other condition deemed by the PI to interfere with the study or increase risk to the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Tolerability as measured by incidence of side effects on an accelerated TMS sensations and adverse events questionnaire | Each morning before treatment and afternoon after treatment during the 5 days of treatment
  Questionnaire asking about the incidence, frequency, and severity of common TMS-related side effects such as headache, tinnitus, and neck pain.
  Higher severity and frequency of side effects indicates lower tolerability
Feasibility as measured by number of the 50 treatments completed | Throughout the 5 days of treatment
  0-50 treatments more treatments completed: higher feasibility

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Before treatment and two weeks after treatment ends
  Depression severity rating scale (0-60, higher numbers indicate higher severity)
Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision, Level 1 Self-Rated Cross-Cutting Symptom Measure (DSM-5-XC) | Before treatment, two weeks after treatment ends, and 3, 6, 9, and 12 months after treatment
  Transdiagnostic rating scale (each question rated 0-4) Minimum score: 0 Maximum score: 92 Higher score indicates worse outcome or worse overall psychiatric burden
World Health Organization Disability Assessment Schedule II (WHODAS 2.0) | Before treatment, two weeks after treatment ends, and 3, 6, 9, and 12 months after treatment
  36-item functional assessment (each question rated 1-5) Minimum: 36 Maximum: 180 Can also be scored by percentiles Higher score indicates more disability

OTHER OUTCOMES:
Beck Depression Inventory (BDI) | Before treatment, daily throughout treatment, two weeks after treatment ends, and 3, 6, 9, and 12 months after treatment
  Depression severity rating scales (0-63, higher numbers indicate higher severity)
Beck Anxiety Inventory (BAI) | Before treatment, daily throughout treatment and two weeks after treatment ends, and 3, 6, 9, and 12 months after treatment
  Anxiety severity rating scale (0-63, higher numbers indicate higher severity)
Adult Attention Deficit/Hyperactivity Disorder Self-Report Scale (AARS) | Before treatment and two weeks after treatment
  ADHD rating scale (each question rated 1-5)
Clinical Global Impression Scale (CGI) | Before treatment and two weeks after treatment
  Global assessment of current symptoms, behavior, and function (1-7)
Illness Intrusiveness Rating Scale (IIRS) | Before treatment, two weeks after treatment, and 3, 6, 9, and 12 months after treatment
  13 item scale measuring how illness affects function. Scored 13-91, higher score indicates higher illness intrusiveness severity
Positive and Negative Symptom Scale (PANSS) | Before treatment and two weeks after treatment
  14 item scale that measures positive and negative symptoms of psychotic disorders. Each question is scored 1-7. Each subscale (positive and negative) is scored 7-49, or total PANSS is scored 14-98. Higher scores indicate greater severity of psychotic symptoms.
Post Traumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Before treatment and two weeks after treatment
  20 item PTSD scale, scored 0-80, higher scores indicate worse symptoms
Yale Brown Obsessive-Compulsive Scale (Y-BOCS) | Before treatment and two weeks after treatment
  OCD assessment tool scored 0-40, higher scores indicate worse outcomes
Emotional Conflict Resolution Test | Before treatment and two weeks after treatment
  Computer task measuring accuracy and reaction time to emotional faces
Learning, Multi-Source Interference Task (MSIT) | Before treatment and two weeks after treatment
  Computer task measuring accuracy and reaction time
Penn Emotion Recognition Task (ER-40) | Before treatment and two weeks after treatment
  Computer task measuring accuracy and reaction time to emotional faces
Death Suicide IAT | Before treatment and two weeks after treatment
  Computer task measuring reaction time
Young Mania Rating Scale (YMRS) | before treatment, daily during treatment, and two weeks after treatment
  11 item scale evaluating mania. Scored 0-60. Higher score indicates worse outcome/higher mania
Hierarchical Taxonomy of Psychopathology Self-Report (HiTOP-SR) | Before treatment and two weeks after treatment
  405-item questionnaire with 87 subspanning a range of psychiatric symptoms. Each item is scored 1-4 (1 = "not at all", 4 = "a lot") and asks whether the following statement has applied to the participant in the past 12 months. Higher scores within any of the 87 sub-scales indicate higher prevalence of that symptom class.
Self-Compassion Scale | Before treatment and two weeks after treatment
  26-item scale (each question rated 1-5). Higher scores indicate less self-compassion

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Taylor, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided